CLINICAL TRIAL: NCT05598112
Title: Effect of Fecal Microbiota Transplantation on Aging and the Underlying Mechanism of Gut Microbiome Restoration: a Randomized Clinical Trial
Brief Title: Effect of Gut Microbiome Intervention on Aging Via Oral FMT
Acronym: STEP-aging
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, Director, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-1784
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Aging; Frailty
Keywords: Aging; Frailty; Microbiome; Treatment; Fecal Microbiota Transplantation
MeSH Terms: conditions — Frailty | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT capsules (Experimental): FMT capsules containing extensively screened donor stool. FMT capsules will be orally taken on week 0, week 4, week 8, week 12, week 24, week 28, week 32, week 36, week 48, week 52, week 56, week 60, week 72, week 76, week 80, week 84.
  Interventions: Biological: FMT capsules
- Placebo capsules (Placebo Comparator): Placebo capsules that do not contain donor stool or any active drug. Placebo capsules will be orally taken on week 0, week 4, week 8, week 12, week 24, week 28, week 32, week 36, week 48, week 52, week 56, week 60, week 72, week 76, week 80, week 84.
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Biological: FMT capsules — FMT capsules containing extensively screened donor stool.
  Arms: FMT capsules
Other: Placebo capsules — Placebo capsules that do not contain donor stool or any active drug.
  Arms: Placebo capsules

SUMMARY:
A severe public health issue facing global population is aging. Increasing preclinical and clinical data indicate the contribution of gut microbiome on aging and aging-related diseases such as cardiovascular disease, Alzheimer Disease, and diabetes. Interventions on microbiota are developed including prebiotics, probiotics, and fecal microbial transplantation (FMT). FMT via oral capsules also advances in recent with limited safety concerns compared with invasive routes. A hypothesis is thus raised that gut microbiome intervention via oral FMT can be a potential safe approach to encourage healthy aging, with multiple aspects evaluated for clinical phenotype of frailty, anthropometric measurement, cognitive function, cardiovascular aging, physical function, living activity, hippocampal volume, telomere length, cognitive biomarkers, inflammatory biomarkers, altered microbial composition and metabolites.

DETAILED DESCRIPTION:
Objective: To explore the effect, safety and underlying mechanisms of gut microbiome intervention via FMT on aging. Study Design: A multi-center, randomized, blinded, placebo-controlled pilot study. Data quality control and statistical analysis: The investigators have invited professional statistic analysts to assist analyzing data and a third party to supervise data quality. Ethics: The Ethics Committee of Fuwai Hospital approved this study. Informed consents before patient enrollment are required.

ELIGIBILITY:
Inclusion Criteria:

1. Age 70-85 years.
2. Patients with informed consent after thorough explanation.

Exclusion Criteria:

1. Participants of other clinical trials;
2. Antibiotics or probiotics usage within last 4 weeks;
3. Severe hepatic or renal diseases ((ALT >3 times the upper limit of normal value, or end stage renal disease on dialysis or eGFR <30 mL/min/1.73 m2, or serum creatinine >2.5 mg/dl [>221 μmol/L]);
4. History of large atherosclerotic cerebral infarction or hemorrhagic stroke (not including lacunar infarction and transient ischemic attack [TIA]);
5. Hospitalization for myocardial infarction within last 6 months; Coronary revascularization (PCI or CABG) within last 12 months; Planned for PCI or CABG in the next 6 months;
6. NYHA class III-IV heart failure; Hospitalization for chronic heart failure exacerbation within last 6 months;
7. Severe valvular diseases; Potential for surgery or percutaneous valve replacement within the study period;
8. Dilated cardiomyopathy; Hypertrophic cardiomyopathy; Rheumatic heart disease; Congenital heart disease;
9. History of dementia, Parkinson's disease, intracranial infection, intracranial tumor, schizophrenia, anxiety, depression;
10. History of neurosurgical operation;
11. History of gastrointestinal tumor, gastrointestinal surgery, inflammatory bowel disease; Hospitalization for peptic ulcer disease exacerbation within last 6 months or anticipated hospitalization for peptic ulcer disease the next 6 months;
12. Hypertension with uncontrolled blood pressure ≥180/110mmHg;
13. Diabetes Mellitus with uncontrolled fasting glucose level ≥200mg/dl (11.1mmol/L), or HbA1C>8%;
14. Addicted to alcohol; Use of medication influencing cognitive function(i.e., antihistamine, antipsychotic);
15. General anesthesia within last 3 months;
16. Other severe diseases influencing the entry or survival of participants, such as malignant tumor or acquired immune deficiency syndrome, life expectancy <1 year;
17. Impaired verbal communication who are incapable of providing their own informed consent, or incapable of self-care;
18. Special diet influencing microbiota (i.e. vegetarian);
19. Other conditions inappropriate for recruitment according to the investigators.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with reduced frailty score at week 96 follow-up | week 96
  Frailty score via CHS criteria of five frailty components, compared with baseline

SECONDARY OUTCOMES:
Proportion of participants with reduced frailty score at week 12 follow-up | week 12
  Frailty score via CHS criteria of five frailty components, compared with baseline
Proportion of participants with reduced frailty score at week 24 follow-up | week 24
  Frailty score via CHS criteria of five frailty components, compared with baseline
Proportion of participants with reduced frailty score at week 48 follow-up | week 48
  Frailty score via CHS criteria of five frailty components, compared with baseline
Proportion of participants with reduced frailty score at week 72 follow-up | week 72
  Frailty score via CHS criteria of five frailty components, compared with baseline
Change from baseline in Frailty score | week 12, week 24, week 48, week 72, week 96, compared with baseline
  Frailty score via CHS criteria of five frailty components, ranging from 0 to 5, with higher score indicating worse outcome
Change from baseline in telomere length | week 48, week 96
  Change from baseline in telomere length
Change from baseline in Cognitive assessment via Mini Mental State Examination(MMSE) | week 24, week 48, week 72, week 96, compared with baseline
  MMSE (Mini Mental State Examination) ranging from 0 to 30, with lower score indicating worse outcome
Change from baseline in Cognitive assessment via Montreal Cognitive Assessment(MoCA) | week 24, week 48, week 72, week 96, compared with baseline
  MoCA (Montreal Cognitive Assessment) ranging from 0 to 30, with lower score indicating worse outcome
Change from baseline in Hippocampal volumes | week 48, week 96
  Hippocampal volumes evaluated by Magnet Resonance Imaging
Change from baseline in cognitive biomarkers | week 12, week 24, week 48, week 72, week 96
  plasma levels of cognitive biomarkers for BDNF、tau、Aβ-40、Aβ42
Change from baseline in inflammatory biomarkers | week 12, week 24, week 48, week 72, week 96
  plasma levels of inflammatory biomarkers for hs-C-reactive protein (hs-CRP)、 interleukin 6(IL-6)、interleukin 1 β(IL-1 β) 、interleukin10 (IL-10)、tumor necrosis factor α(TNF-α)
Change from baseline in Intestinal Microbiota Composition Pre- and Post-intervention via Metagenomic Analysis | week 12, week 24, week 48, week 72, week 96
  Change in Intestinal Microbiota Composition Pre- and Post-intervention (FMT or Placebo) via Metagenomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Change from baseline in Intestinal Microbiota Function assessed by KEGG Orthology (KO) Pre- and Post-intervention via Metagenomic Analysis | week 12, week 24, week 48, week 72, week 96
  Change in Intestinal Microbiota Function assessed by KEGG Orthology (KO) Pre- and Post-intervention (FMT or Placebo) via Metagenomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Change from baseline in Plasma Metabolite Composition Pre- and Post-intervention via Metabolomic Analysis | week 12, week 24, week 48, week 72, week 96
  Change in Plasma Metabolite Composition Pre-and Post-intervention (FMT or Placebo) via Metabolomic Analysis
Change from baseline in Ankle-Brachial Blood Pressure Index(ABI) | week 48, week 96
  Change for ABI as an objective measurement of arterial insufficiency based on the ratio of ankle systolic pressure to brachial systolic pressure.
Change from baseline in Pulse wave velocity(PWV) | week 48, week 96
  Change for Pulse wave velocity(PWV)
Number of Participants with Adverse Events (AEs) as a Measure of Safety | week 12, week 24, week 48, week 72, week 96
  Number of Participants with Adverse Events (AEs) as a Measure of Safety
Change from baseline in Body Mass Index (BMI) | week 4, week 8, week 12, week 24, week 48, week 72, week 96
  Change for Body Mass Index
Change from baseline in office SBP | week 4, week 8, week 12, week 24, week 48, week 72, week 96
  change for office systolic blood pressure(SBP)
Change from baseline in office DBP | week 4, week 8, week 12, week 24, week 48, week 72, week 96
  change for office diastolic blood pressure(DBP)
Change from baseline in Blood Lipid Level | week 12, week 24, week 48, week 96
  Change for Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol)
Change from baseline in blood fasting glucose level | week 12, week 24, week 48, week 96
  Change for blood fasting glucose level
Change from baseline in blood HbA1c level | week 12, week 24, week 48, week 96
  Change for blood glycosylated hemoglobin, type A1C (HbA1c) level
Change from baseline in physical function assessment via 6MWT | week 12, week 24, week 48, week 72, week 96
  6-minute walking test(6MWT)
Change from baseline in daily function assessment via Activity of Daily Living (ADL) | week 12, week 24, week 48, week 72, week 96
  Activity of Daily Living (ADL) ranging from 0 to 100, with lower score indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD,PhD, Principal Investigator — Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart, Lung and Blood Vessel Diseases, Chinese Institutes for Medical Research
Locations (6):
- China (6):
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The collected data, study protocol, and SAP are planned to be shared after the study ends 3 years later (anticipated)
Supporting Information: Study Protocol, SAP
Time Frame: after the study ends 3 years later (anticipated)
Access Criteria: Access to these deidentified data will be required for written permission from the responsible investigation center and only for qualified researchers.

REFERENCES:
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Ghosh TS, Rampelli S, Jeffery IB, Santoro A, Neto M, Capri M, Giampieri E, Jennings A, Candela M, Turroni S, Zoetendal EG, Hermes GDA, Elodie C, Meunier N, Brugere CM, Pujos-Guillot E, Berendsen AM, De Groot LCPGM, Feskins EJM, Kaluza J, Pietruszka B, Bielak MJ, Comte B, Maijo-Ferre M, Nicoletti C, De Vos WM, Fairweather-Tait S, Cassidy A, Brigidi P, Franceschi C, O'Toole PW. Mediterranean diet intervention alters the gut microbiome in older people reducing frailty and improving health status: the NU-AGE 1-year dietary intervention across five European countries. Gut. 2020 Jul;69(7):1218-1228. doi: 10.1136/gutjnl-2019-319654. Epub 2020 Feb 17. PMID 32066625
- [Result] Ng TP, Feng L, Nyunt MS, Feng L, Niti M, Tan BY, Chan G, Khoo SA, Chan SM, Yap P, Yap KB. Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal Among Older Adults: A Randomized Controlled Trial. Am J Med. 2015 Nov;128(11):1225-1236.e1. doi: 10.1016/j.amjmed.2015.06.017. Epub 2015 Jul 6. PMID 26159634
- [Result] Mullish BH, Quraishi MN, Segal JP, McCune VL, Baxter M, Marsden GL, Moore DJ, Colville A, Bhala N, Iqbal TH, Settle C, Kontkowski G, Hart AL, Hawkey PM, Goldenberg SD, Williams HRT. The use of faecal microbiota transplant as treatment for recurrent or refractory Clostridium difficile infection and other potential indications: joint British Society of Gastroenterology (BSG) and Healthcare Infection Society (HIS) guidelines. Gut. 2018 Nov;67(11):1920-1941. doi: 10.1136/gutjnl-2018-316818. Epub 2018 Aug 28. PMID 30154172
- [Result] Kundu P, Lee HU, Garcia-Perez I, Tay EXY, Kim H, Faylon LE, Martin KA, Purbojati R, Drautz-Moses DI, Ghosh S, Nicholson JK, Schuster S, Holmes E, Pettersson S. Neurogenesis and prolongevity signaling in young germ-free mice transplanted with the gut microbiota of old mice. Sci Transl Med. 2019 Nov 13;11(518):eaau4760. doi: 10.1126/scitranslmed.aau4760. PMID 31723038